CLINICAL TRIAL: NCT00478231
Title: A Multicenter, Open Label, Non-Comparative Safety Study Of Maraviroc
Brief Title: Multicenter, Safety Study Of Maraviroc
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4001063
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Results first posted 2011-08-08 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infection
Keywords: Multicenter; Open Label; Non-Comparative Safety Study Of Maraviroc; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Maraviroc should be dosed BID with total dose adjusted according to the other drugs the patient is taking. Maraviroc may be taken with or without food. The subject should only take missed doses if it is not within 6 hours prior to the planned next dose. No dose adjustment of OBT is required due to the presence of maraviroc.

SUMMARY:
To collect safety and tolerability data in a more diverse patient population of patients with HIV/Aids, who have limited therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with limited or no approved treatment options available to them due to resistance or intolerance;
* Subjects must be failing to achieve adequate virologic suppression on their current regimen and have HIV-1 RNA ≥ 1000 copies/ml, at screening.
* Have only R5 HIV-1 at Screening as verified by the Monogram Biosciences Trofile assay.

Exclusion Criteria:

* Failed prior treatment with any CCR5 antagonist, in any ongoing CCR5 trials or having previously discontinued Maraviroc in trials
* Potentially life threatening (Grade 4) laboratory abnormality or medical condition (according to the Division of AIDS table for grading severity of adult adverse experiences) still under investigation unless a diagnosis has been established and felt not to affect risk/benefit assessment or eventual interpretation of safety results, based on discussion between the investigator and Pfizer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2007-07; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- Brazil (11):
  - Pfizer Investigational Site, Salvador, Estado de Bahia
  - Pfizer Investigational Site, Brasília, Federal District
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Nova Iguaçu, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Florianópolis, Santa Catarina
  - Pfizer Investigational Site, Campinas, São Paulo
  - Pfizer Investigational Site, Ribeirão Preto, São Paulo
  - Pfizer Investigational Site, Santo André, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo

REFERENCES:
- [Derived] Furtado J, Madruga JV, Bicudo EL, da Eira M, Lopes MI, Netto EM, Santini-Oliveira M, Leite OH, Machado AA, Tupinambas U, de Andrade Neto JL, Lima MP, Pedro Rde J, Miranda AF, Lewi DS, Santos BR, Portsmouth S, Wajsbrot DB, Cassoli LM. Safety and immunovirologic outcomes with maraviroc combination regimens in patients with a history of past treatment failures and virologic resistance in Brazil: an open-label, multicenter phase 3b study. AIDS Res Hum Retroviruses. 2013 Sep;29(9):1203-10. doi: 10.1089/AID.2012.0330. Epub 2013 Jun 25. PMID 23731330
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001063&StudyName=Multicenter%2C%20Safety%20Study%20Of%20Maraviroc

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 638 participants were screened, out of which 429 participants were screen failures and 209 were assigned to the study treatment.
Groups:
- Maraviroc: Maraviroc tablet 150 to 600 milligrams (mg) twice daily (BID), dose adjusted according to the other prescribed drugs taken by participants as part of optimized background therapy (OBT) selected according to local standard of care.
Period: Overall Study
Arm/Group | Maraviroc
Started | 209
Treated | 206
Completed | 125
Not Completed | 84
Not completed — Death | 7
Not completed — Lack of Efficacy | 47
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 6
Not completed — Other | 9
Not completed — Adverse Event | 5
Not completed — Randomized, not treated | 3

BASELINE CHARACTERISTICS:
Arm/Group | Maraviroc
Number analyzed (Participants) | 206
Age Continuous [Mean (Standard Deviation); unit: Years] | 43.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 145

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 and Grade 4 Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AEs: any untoward medical occurrence/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was congenital anomaly. Grade 3: Events that interrupted participant's usual daily activity and traditionally required systemic drug therapy or other treatment. Grade 4: Events which were unacceptable and intolerable or which were irreversible or caused participant to be in imminent danger of death.
Time Frame: Baseline to 30 days post-week 96 or early termination (ET)
Population: The safety analysis set composed of all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 206
Participants
  Grade 3 AEs | 40
  Grade 4 AEs | 9
  SAEs | 34

2. Primary Outcome: Number of Participants With Division of Acquired Immunodeficiency Syndrome (DAIDS) Grade 3 and Grade 4 Laboratory Abnormalities
Description: Grade 3 or severe events included those that interrupted participant's usual daily activity and traditionally required systemic drug therapy or other treatment. Grade 4 or very severe events included those that were unacceptable and intolerable or which were irreversible or caused the participant to be in imminent danger of death.
Time Frame: Baseline to 30 days post-week 96 or ET
Population: The safety analysis set composed of all participants who received at least one dose of study medication. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the time point for each group respectively.
Measure: Number; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 206
Participants
  Grade 3: Alanine aminotransferase (ALT) | 0
  Grade 3: Aspartate aminotransferase (AST) | 4
  Grade 3: Absolute neutrophil count (ANC) | 7
  Grade 3: Alkaline phosphatase | 1
  Grade 3: Gamma-glutamyl transpeptidase (GGT) | 15
  Grade 3: Hyperbilirubinemia | 17
  Grade 3: Hyperuricemia | 3
  Grade 3: Lipase (n= 101) | 8
  Grade 3: Platelets | 3
  Grade 3: Potassium (Hyperkalemia) | 0
  Grade 3: Serum amylase | 12
  Grade 4: Alanine aminotransferase (ALT) | 1
  Grade 4: Aspartate aminotransferase (AST) | 0
  Grade 4: Absolute neutrophil count (ANC) | 4
  Grade 4: Alkaline phosphatase | 0
  Grade 4: Gamma-glutamyl transpeptidase (GGT) | 8
  Grade 4: Hyperbilirubinemia | 6
  Grade 4: Hyperuricemia | 1
  Grade 4: Lipase (n= 101) | 2
  Grade 4: Platelets | 0
  Grade 4: Potassium (Hyperkalemia) | 2
  Grade 4: Serum amylase | 1

3. Primary Outcome: Number of Participants With Treatment Emergent Malignancies
Time Frame: Baseline to 30 days post-week 96 or ET
Population: The safety analysis set composed of all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 206
Participants
  Carcinoma in situ | 1
  Hodgkin's disease | 1
  Intestinal T-cell lymphoma | 1
  Neoplasm of appendix | 1

4. Primary Outcome: Number of Participants With Category C Acquired Immunodeficiency Syndrome (AIDS) Related Infections
Description: Number of participants with AIDS-related infections based on investigator classification guided by a predefined list of clinical Category C AEs per Center for Disease Control (CDC) HIV Classification System.
Time Frame: Baseline to 30 days post-week 96 or ET
Population: The safety analysis set composed of all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 206
Participants
  Cerebral toxoplasmosis | 2
  Disseminated cryptococcosis | 1
  Oesophageal candidiasis | 3
  Pneumocystis jiroveci pneumonia | 3
  Leukoencephalopathy | 1

5. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Pre-defined criteria based on upper limit normal (ULN) and lower limit normal (LLN) were established for each laboratory test to define the values that would be identified as laboratory test abnormality.
Time Frame: Baseline to 30 days post-week 96 or ET
Population: The safety analysis set composed of all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 206
Participants
  Hematocrit (<0.8*LLN) | 13
  Red blood cell count (<0.8*LLN) | 35
  White blood cell count (<0.6*LLN) | 7
  White blood cell count (>1.5*ULN) | 4
  Absolute lymphocytes (<0.8*LLN) | 12
  Absolute lymphocytes (>1.2*ULN) | 60
  Percent lymphocytes (<0.8*LLN) (n= 1) | 0
  Percent lymphocytes (>1.2*ULN) (n= 1) | 1
  Percent neutrophils (<0.8*LLN) (n= 1) | 1
  Percent neutrophils (>1.2*ULN) (n= 1) | 0
  Absolute basophils (>1.2*ULN) | 10
  Percent basophils (>1.2*ULN) (n= 1) | 0
  Absolute eosinophils (>1.2*ULN) | 32
  Percent eosinophils (>1.2*ULN) (n= 1) | 0
  Absolute monocytes (>1.2*ULN) | 25
  Percent monocytes (>1.2*ULN) (n= 1) | 0
  Direct Bilirubin (>1.5*ULN) | 67
  Indirect bilirubin (>1.5*ULN) | 25
  Lactose dehydrogenase (LDH) (>3.0*ULN) | 1
  Total protein (<0.8*LLN) | 1
  Total protein (>1.2*ULN) | 19
  Albumin (<0.8*LLN) | 3
  Albumin (>1.2*ULN) | 0
  Blood urea nitrogen (BUN) (>1.3*ULN) | 7
  Cholesterol (>1.3*ULN) | 26
  High density lipoprotein cholesterol (<0.8*LLN) | 115
  Low density lipoprotein cholesterol (>1.2*ULN) | 101
  Triglycerides (>1.3*ULN) | 145
  Calcium (<0.9*LLN) | 6
  Calcium (>1.1*ULN) | 0
  Creatine kinase (CK) (>2.0*ULN) | 50

6. Secondary Outcome: Percentage of Participants With at Least 0.5 Log 10 Reduction in Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA)
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84 and Week 96 or end of treatment (EOT)
Population: The full analysis set (FAS) included all participants who had taken at least one dose of study drug and provided any post-baseline efficacy evaluation. The 'n' signifies those participants who received study drug and were evaluated for this measure at time point for each group respectively. Last Observation Carried Forward (LOCF) method was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 206
Percentage of participants
  Week 4 (n= 202) | 78.7
  Week 8 (n= 196) | 78.6
  Week 12 (n= 190) | 80.5
  Week 24 (n= 185) | 79.5
  Week 36 (n= 171) | 83.6
  Week 48 (n= 158) | 82.3
  Week 60 (n= 141) | 84.4
  Week 72 (n= 137) | 81.0
  Week 84 (n= 125) | 82.4
  Week 96 or EOT (n= 109) | 89.9
  LOCF (n= 206) | 76.2

7. Secondary Outcome: Percentage of Participants With at Least 1.0 Log 10 Reduction in HIV-1 RNA
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84 and Week 96 or EOT
Population: The FAS included all the participants who had taken at least one dose of the study drug and provided any post-baseline efficacy evaluation. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the time point for each group respectively. Missing data was imputed using LOCF.
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 206
Percentage of participants
  Week 4 (n= 202) | 67.8
  Week 8 (n= 196) | 68.9
  Week 12 (n= 190) | 71.1
  Week 24 (n= 185) | 68.6
  Week 36 (n= 171) | 69.0
  Week 48 (n= 158) | 70.3
  Week 60 (n= 141) | 70.2
  Week 72 (n= 137) | 64.2
  Week 84 (n= 125) | 71.2
  Week 96 or EOT (n= 109) | 72.5
  LOCF (n= 206) | 61.2

8. Secondary Outcome: Percentage of Participants Achieving HIV-1 RNA Below Limit of Quantification
Description: Below limit of quantification was defined as less than 400 copies/milliliter (mL)
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84 and Week 96 or EOT
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 206
Percentage of participants
  Baseline | 2.4
  Week 4 (n= 202) | 29.7
  Week 8 (n= 196) | 43.9
  Week 12 (n= 190) | 42.6
  Week 24 (n= 185) | 41.1
  Week 36 (n= 171) | 47.4
  Week 48 (n= 158) | 41.1
  Week 60 (n= 141) | 36.2
  Week 72 (n= 137) | 24.8
  Week 84 (n= 125) | 23.2
  Week 96 or EOT (n= 109) | 33.9
  LOCF (n= 206) | 26.7

9. Secondary Outcome: Change From Baseline in Lymphocyte Cluster of Differentiation 4 (CD4) Count at Week 4, 8, 12, 24, 36, 48, 60, 72, 84 and Week 96 or EOT
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84 and Week 96 or EOT
Population: The FAS population included all the participants who had taken at least one dose of the study drug and provided any post-baseline efficacy evaluation. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the time point for each group respectively. Missing data was imputed using LOCF.
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/µL)
Arm/Group | Maraviroc
Number analyzed (Participants) | 202
cells per microliter (cells/µL)
  Baseline | 215.6 (179.9)
  Change at Week 4 (n= 190) | 93.5 (96.7)
  Change at Week 8 (n= 190) | 110.0 (95.2)
  Change at Week 12 (n= 186) | 132.1 (164.1)
  Change at Week 24 (n= 184) | 137.3 (115.0)
  Change at Week 36 (n= 165) | 157.8 (128.4)
  Change at Week 48 (n= 154) | 172.2 (124.0)
  Change at Week 60 (n= 134) | 187.2 (140.4)
  Change at Week 72 (n= 129) | 199.8 (161.0)
  Change at Week 84 (n= 124) | 198.2 (177.3)
  Change at Week 96 or EOT (n= 107) | 225.2 (175.3)
  Change at LOCF (n= 201) | 174.1 (168.5)

10. Secondary Outcome: Change From Baseline in Lymphocyte Cluster of Differentiation 8 (CD8) Count at Week 4, 8, 12, 24, 36, 48, 60, 72, 84 and Week 96 or EOT
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84 and Week 96 or EOT
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Maraviroc
Number analyzed (Participants) | 202
cells/µL
  Baseline | 1016.4 (676.3)
  Change at Week 4 (n= 190) | 387.3 (597.0)
  Change at Week 8 (n= 190) | 518.3 (666.4)
  Change at Week 12 (n= 186) | 507.2 (685.6)
  Change at Week 24 (n= 185) | 358.1 (577.2)
  Change at Week 36 (n= 165) | 352.3 (545.3)
  Change at Week 48 (n= 155) | 348.6 (591.0)
  Change at Week 60 (n= 135) | 349.1 (566.7)
  Change at Week 72 (n= 130) | 272.4 (594.8)
  Change at Week 84 (n= 124) | 246.7 (567.3)
  Change at Week 96 or EOT (n= 107) | 214.5 (593.2)
  Change at LOCF (n= 201) | 223.0 (562.0)

11. Secondary Outcome: Change From Baseline in CD4 Percent at Week 4, 8, 12, 24, 36, 48, 60, 72, 84 and Week 96 or EOT
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84 and Week 96 or EOT
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent CD4
Arm/Group | Maraviroc
Number analyzed (Participants) | 202
Percent CD4
  Baseline | 12.2 (7.5)
  Change at Week 4 (n= 190) | 1.8 (3.4)
  Change at Week 8 (n= 190) | 1.3 (3.2)
  Change at Week 12 (n= 186) | 2.1 (4.4)
  Change at Week 24 (n= 184) | 2.9 (3.7)
  Change at Week 36 (n= 165) | 3.6 (3.9)
  Change at Week 48 (n= 154) | 4.3 (4.1)
  Change at Week 60 (n= 134) | 4.5 (4.5)
  Change at Week 72 (n= 129) | 5.2 (4.3)
  Change at Week 84 (n= 124) | 5.3 (5.2)
  Change at Week 96 or EOT (n= 107) | 6.6 (5.1)
  Change at LOCF (n= 201) | 4.9 (5.3)

12. Secondary Outcome: Change From Baseline in CD8 Percent at Week 4, 8, 12, 24, 36, 48, 60, 72, 84 and Week 96 or EOT
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84 and Week 96 or EOT
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent CD8
Arm/Group | Maraviroc
Number analyzed (Participants) | 202
Percent CD8
  Baseline | 59.8 (13.1)
  Change at Week 4 (n= 190) | 0.4 (6.1)
  Change at Week 8 (n= 190) | 0.9 (7.3)
  Change at Week 12 (n= 186) | -0.1 (8.2)
  Change at Week 24 (n= 185) | -2.5 (8.3)
  Change at Week 36 (n= 165) | -3.6 (8.6)
  Change at Week 48 (n= 155) | -4.3 (9.9)
  Change at Week 60 (n= 135) | -4.7 (10.4)
  Change at Week 72 (n= 130) | -6.1 (10.9)
  Change at Week 84 (n= 124) | -6.8 (10.3)
  Change at Week 96 or EOT (n= 107) | -7.7 (10.7)
  Change at LOCF (n= 201) | -5.4 (10.6)

13. Secondary Outcome: Number of Participants With C-X-C Chemokine Receptor Type 4 {CXCR4} [X4] Tropism Status
Description: Virus tropism was done by the Monogram Biosciences Trofile assay.
Time Frame: Time of virologic failure (VF) and Week 96 or EOT
Population: The FAS included all the participants who had taken at least one dose of the study drug and provided any post-baseline efficacy evaluation. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the time point for each group respectively.
Measure: Number; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 206
Participants
  VF X4 (n= 134) | 7
  EOT X4 (n= 146) | 8

14. Other Pre Specified Outcome: Change From Baseline in Human Immunodeficiency Virus (HIV) -1 Viral Load (Ribonucleic Acid [RNA]) at Week 4, 8, 12, 24, 36, 48, 60, 72, 84 and Week 96 or EOT
Description: Change from baseline in log 10-transformed plasma viral load (HIV-1 RNA) levels (log 10 copies per milliliter [log10 copies/ml]).
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84 and Week 96 or EOT
Population: The FAS included all participants who had taken at least one dose of study drug and provided any post-baseline efficacy evaluation. The 'n' signifies those participants who received study drug and were evaluated for this measure at time point for each group respectively. Missing data was imputed using LOCF.
Measure: Mean (Standard Deviation); unit: log 10 copies/ml
Arm/Group | Maraviroc
Number analyzed (Participants) | 206
log 10 copies/ml
  Baseline | 4.8 (0.9)
  Change at week 4 (n= 202) | -1.5 (1.0)
  Change at week 8 (n= 196) | -1.5 (1.1)
  Change at week 12 (n= 190) | -1.6 (1.1)
  Change at week 24 (n= 185) | -1.6 (1.1)
  Change at week 36 (n= 171) | -1.6 (1.0)
  Change at week 48 (n= 158) | -1.6 (1.0)
  Change at week 60 (n= 141) | -1.6 (1.1)
  Change at week 72 (n= 137) | -1.4 (1.1)
  Change at week 84 (n= 125) | -1.5 (1.1)
  Change at week 96 or EOT (n= 109) | -1.7 (1.0)
  Change at LOCF (n= 206) | -1.4 (1.1)

15. Other Pre Specified Outcome: Time to Virologic Failure (VF)
Description: Virologic failure was defined as failing to achieve a reduction in HIV-1 RNA of at least 0.5 log10 copies/ml from baseline by the second viral load determination; or experiencing at least 0.5 log10 increase from nadir in HIV-1 RNA after achieving an HIV-1 RNA reduction from baseline more than 0.5 log10 copies/ml; or experiencing an HIV-1 RNA more than 1000 copies/ml after having achieved an HIV-1 RNA below level of quantification.
Time Frame: Baseline to Week 96 or EOT
Population: The FAS included all the participants who had taken at least one dose of the study drug and provided any post-baseline efficacy evaluation.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Maraviroc
Number analyzed (Participants) | 206
Days | 255.0 [172.0 to 336.0]

16. Other Pre Specified Outcome: Number of Participants With Genotype Resistance
Description: Evolution in resistance to OBT was shown by emergence of new primary or secondary resistance mutations to nucleoside reverse transcriptase inhibitor (NRTI), non-nucleoside reverse transcriptase inhibitor (NNRTI) and protease inhibitor (PI).
Time Frame: Baseline through Week 96
Population: FAS included all the participants who had taken at least one dose of the study drug and provided any post-baseline efficacy evaluation. Here, the 'N = 167' is signifying those participants who were evaluable for this measure at the specified time point for this arm group.
Measure: Number; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 167
Participants
  VF: NRTI | 0
  VF: NNRTI | 0
  VF: PI | 16
  VF: NRTI and NNRTI | 0
  VF: NRTI and PI | 32
  VF: NNRTI and PI | 7
  VF: NRTI and NNRTI and PI | 64
  VF: no NRTI, no NNRTI and no PI | 0
  VF: no test result data | 48

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Maraviroc
Serious Adverse Events (participants affected / at risk) | 34/206
Other Adverse Events (participants affected / at risk) | 185/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc (N=206)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Anal fistula (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Fat tissue increased (General disorders) | 1
Gait disturbance (General disorders) | 1
Pyrexia (General disorders) | 3
Hepatitis (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Cerebral toxoplasmosis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Disseminated cryptococcosis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Keratitis herpetic (Infections and infestations) | 1
Meningitis meningococcal (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 4
Muscle rupture (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Blood bilirubin increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intestinal T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pseudomyxoma peritonei (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urethral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 3
Guillain-Barre syndrome (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Monoplegia (Nervous system disorders) | 1
Optic neuritis (Nervous system disorders) | 1
Bradyphrenia (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Victim of homicide (Social circumstances) | 1
Haematoma (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc (N=206)
Anaemia (Blood and lymphatic system disorders) | 8
Eosinophilia (Blood and lymphatic system disorders) | 2
Granulocytopenia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 9
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Arrhythmia (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Cleft lip (Congenital, familial and genetic disorders) | 1
Congenital optic nerve anomaly (Congenital, familial and genetic disorders) | 1
Porphyria non-acute (Congenital, familial and genetic disorders) | 1
Ear disorder (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Hypoacusis (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Vestibular disorder (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Conjunctival hyperaemia (Eye disorders) | 2
Conjunctivitis (Eye disorders) | 2
Conjunctivitis allergic (Eye disorders) | 1
Dacryostenosis acquired (Eye disorders) | 1
Eye disorder (Eye disorders) | 1
Eye pain (Eye disorders) | 2
Eye pruritus (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 5
Ocular icterus (Eye disorders) | 4
Ulcerative keratitis (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 11
Aerophagia (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Anal haemorrhage (Gastrointestinal disorders) | 1
Anal ulcer (Gastrointestinal disorders) | 1
Breath odour (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 10
Dental necrosis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 33
Dry mouth (Gastrointestinal disorders) | 2
Duodenitis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 8
Food poisoning (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastric disorder (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 5
Hiatus hernia (Gastrointestinal disorders) | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Leukoplakia oral (Gastrointestinal disorders) | 1
Lip oedema (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 17
Odynophagia (Gastrointestinal disorders) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Rectal discharge (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 14
Administration site pain (General disorders) | 1
Adverse drug reaction (General disorders) | 1
Application site nodule (General disorders) | 3
Application site pain (General disorders) | 2
Asthenia (General disorders) | 8
Chest pain (General disorders) | 6
Chills (General disorders) | 1
Crepitations (General disorders) | 2
Fatigue (General disorders) | 1
Feeling hot (General disorders) | 2
Gait disturbance (General disorders) | 1
Influenza like illness (General disorders) | 5
Injection site erythema (General disorders) | 1
Injection site nodule (General disorders) | 9
Injection site pain (General disorders) | 1
Injection site reaction (General disorders) | 1
Malaise (General disorders) | 1
Nodule (General disorders) | 2
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 6
Pain (General disorders) | 1
Pyrexia (General disorders) | 9
Ulcer (General disorders) | 1
Xerosis (General disorders) | 2
Hepatic steatosis (Hepatobiliary disorders) | 4
Hepatomegaly (Hepatobiliary disorders) | 2
Hepatosplenomegaly (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Allergy to arthropod bite (Immune system disorders) | 1
Food allergy (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 5
Acarodermatitis (Infections and infestations) | 4
Acute sinusitis (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Anogenital warts (Infections and infestations) | 6
Arthropod infestation (Infections and infestations) | 1
Bacterial diarrhoea (Infections and infestations) | 1
Body tinea (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 2
Bronchitis bacterial (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 3
Cerebral toxoplasmosis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Dental fistula (Infections and infestations) | 1
Dermatophytosis (Infections and infestations) | 3
Ear infection (Infections and infestations) | 2
Erysipelas (Infections and infestations) | 2
Folliculitis (Infections and infestations) | 2
Fungal infection (Infections and infestations) | 1
Furuncle (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 3
Gastrointestinal candidiasis (Infections and infestations) | 1
Genital candidiasis (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 8
HIV infection (Infections and infestations) | 1
Herpes ophthalmic (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 8
Herpes simplex ophthalmic (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 13
Herpes zoster ophthalmic (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 13
Labyrinthitis (Infections and infestations) | 3
Laryngitis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Lymphogranuloma venereum (Infections and infestations) | 1
Molluscum contagiosum (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 32
Necrotising herpetic retinopathy (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 3
Onychomycosis (Infections and infestations) | 6
Oral candidiasis (Infections and infestations) | 8
Oral herpes (Infections and infestations) | 3
Papilloma viral infection (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Parotitis (Infections and infestations) | 2
Pneumocystis jiroveci pneumonia (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 8
Pneumonia bacterial (Infections and infestations) | 4
Pneumonia primary atypical (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 1
Secondary syphilis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 18
Sinusitis bacterial (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 2
Syphilis (Infections and infestations) | 1
Tinea cruris (Infections and infestations) | 2
Tinea pedis (Infections and infestations) | 5
Tinea versicolour (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 4
Tonsillitis bacterial (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 17
Urethritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vaginitis bacterial (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 2
Vulvovaginal candidiasis (Infections and infestations) | 1
Vulvovaginitis (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Chest injury (Injury, poisoning and procedural complications) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 2
Medication error (Injury, poisoning and procedural complications) | 2
Procedural pain (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Scratch (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 5
Blood amylase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 6
Blood creatine phosphokinase increased (Investigations) | 13
Blood creatinine increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Blood testosterone decreased (Investigations) | 1
Blood triglycerides increased (Investigations) | 4
Breath sounds abnormal (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
High density lipoprotein decreased (Investigations) | 7
Lipase increased (Investigations) | 1
Weight decreased (Investigations) | 4
Weight increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 17
Hyperuricaemia (Metabolism and nutrition disorders) | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypovitaminosis (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 4
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anosmia (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 13
Dysaesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 22
Hyperaesthesia (Nervous system disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Monoparesis (Nervous system disorders) | 1
Myoclonus (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 4
Optic neuritis (Nervous system disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 2
Sleep phase rhythm disturbance (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 5
Adjustment disorder with depressed mood (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 11
Disorientation (Psychiatric disorders) | 1
Impatience (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 12
Libido decreased (Psychiatric disorders) | 1
Libido increased (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Stress (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Albuminuria (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 2
Nephropathy (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Breast cyst (Reproductive system and breast disorders) | 1
Breast enlargement (Reproductive system and breast disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 3
Genital lesion (Reproductive system and breast disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 1
Haematospermia (Reproductive system and breast disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Vaginal lesion (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Androgenetic alopecia (Skin and subcutaneous tissue disorders) | 1
Chloasma (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Eosinophilic pustular folliculitis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Facial wasting (Skin and subcutaneous tissue disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Leukoplakia (Skin and subcutaneous tissue disorders) | 1
Lipoatrophy (Skin and subcutaneous tissue disorders) | 2
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 5
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 2
Papule (Skin and subcutaneous tissue disorders) | 2
Prurigo (Skin and subcutaneous tissue disorders) | 14
Pruritus (Skin and subcutaneous tissue disorders) | 11
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 15
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 6
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 22
Urticaria (Skin and subcutaneous tissue disorders) | 1
Urticaria papular (Skin and subcutaneous tissue disorders) | 1
Mass excision (Surgical and medical procedures) | 1
Varicose vein operation (Surgical and medical procedures) | 1
Arteriosclerosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 2
Hyperaemia (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 2
Orthostatic hypotension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.